CLINICAL TRIAL: NCT00194051
Title: Symptomatic, Biomechanical and Radiographic Outcomes in Knee Osteoarthritis Following Gastric Bypass Surgery
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Elizabeth Severance Prentiss Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 02-03-10
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Osteoarthritis
Keywords: obesity; gait biomechanics; knee osteoarthritis
MeSH Terms: conditions — Obesity; Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: gastric bypass surgery

SUMMARY:
Weight is a risk factor for knee osteoarthritis

Knee osteoarthritis is associated with abnormal gait biomechanics

Gait biomechanics are evaluated in gastric bypass patients before and after losing 100 pounds.

DETAILED DESCRIPTION:
Weight is a major risk factor for development of knee osteoarthritis, but not hip or ankle arthritis. One possible mechanism for this is the generation of abnormal gait biomechanics secondary to obesity that are conducive to the development of knee osteoarthritis.

We evaluate gait biomechanics, knee symptoms and knee radiographs in 35 obese patients before and after gastric bypass surgery to determine the effect of significant weight loss on gait biomechanics, knee symptoms and knee radiographs.

ELIGIBILITY:
Inclusion Criteria:

Undergoing gastric bypass surgery At least 35 years old

-

Exclusion Criteria:

Inability to walk unassisted Pain affecting gait in any lower extremity joint

-

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2006-05-01 (Actual); Study Completion 2006-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Hooper, MD, MS, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States